CLINICAL TRIAL: NCT04291625
Title: Evaluation of Intraoperative Lagophthalmos Formula for Levator Resection in Congenital Ptosis on Egyptian Patients
Brief Title: Evaluation of Intraoperative Lagophthalmos Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Sameh S. Mandour, Assistant Professor of Ophthalmology, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19519OPHT38
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Ptosis, Eyelid
Keywords: congenital; ptosis; levator function; MRD 1
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: 20 eyelids with congenital ptosis with levator function of 4 mm or better, who underwent levator muscle resection guided by the recent intraoperative lagophthalmos formula.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- congenital ptosis (Other): children who had congenital ptosis with levator function of 4mm or better, underwent levator muscle resection guided by intraoperative lagophthalmos formula.
  Interventions: Procedure: Levator muscle resection

INTERVENTIONS:
Procedure: Levator muscle resection — Surgery was performed under general anaesthesia. Two milliliters of 2% lidocaine with 1:100 000 epinephrine is injected subcutaneously. After the upper eyelid incision at the desired crease line, the orbital septum was opened and the preaponeurotic fat was identified and dissected off the levator aponeurosis. The aponeurosis was disinserted from the tarsus, and the complex of levator aponeurosis and Muller muscle was dissected free from the conjunctiva. The desired eyelid height was determined from the proposed formula.
  Satisfactory Intraoperative lagophthalmos was defined as a difference of less than 1 mm between recommended by the formula and actual intraoperative lagophthalmos.
  After permanent fixation, a caliper was used for precise measurement of lagophthalmos in a supine position. Additional sutures were placed on the medial and lateral sides for satisfactory eyelid contour. The redundant levator complex was excised. Eyelid crease was made by placing three interrupted sutures

SUMMARY:
This is a prospective non-randomized study to evaluate the recent intraoperative lagophthalmos formula method for levator resection in determining postoperative eyelid height in congenital ptosis on Egyptian children. included 20 eyelids from 17 Egyptian children with congenital ptosis with levator function of 4mm or better, they underwent levator muscle resection guided by the recent intraoperative lagophthalmos formula

DETAILED DESCRIPTION:
This is a prospective non-randomized study to evaluate the recent intraoperative lagophthalmos formula method for levator resection in determining postoperative eyelid height in congenital ptosis on Egyptian children. The study included 20 eyelids of 17 Egyptian children with congenital ptosis with levator function of 4mm or better, they underwent levator muscle resection guided by the recent intraoperative lagophthalmos formula.

Preoperative MRD 1 (Margin-to-reflex distance 1) and levator function were measured, then intraoperative palpebral fissure opening was determined from formula: Intraoperative lagophthalmos=9.08 - 0.48×Preoperative MRD1 - 0.26× Levator function. Postoperative MRD 1 was measured after 1 day, 1week,1month, 3 months and 6 months .Success was defined as postoperative MRD 1 ≥ 3 mm and difference between both eyelids height ≤ 1 mm at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* simple congenital ptosis (any degree) with levator function of 4mm or more

Exclusion Criteria:

* levator function less than 4mm
* a history of previous ptosis surgery
* other accompanying congenital diseases, such as blepharophimosis, congenital fibrosis of the extraocular muscles, Marcus Gunn (jaw-winking) syndrome, double elevator palsy and congenital third nerve palsy

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Chick the validity of Lagophthalmos formula for Egyptian children with congenital ptosis | 6 months
  We apply the following formula:
  Intraoperative lagophthalmos=9.08 - 0.48×Preoperative MRD1 - 0.26×Levator function.
  We tried to achieve the calculated lagophthalmos by the formula intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rakha, MBBch, Study Chair — Kafr Elsheikh eye surgery center, Kafr Elsheikh, Egypt; Amr Awara, MD, Study Chair — Tanta University, Tanta, Gharbia, Egypt; Abdel Khalek I Elsaadany, PhD, Study Director — Menoufia University, Shebin El Koum, Menoufia, Egypt
Locations (1):
- Ophthalmology Department, Menoufia University Hospital, Shibīn al Kawm, Menoufia, Egypt